CLINICAL TRIAL: NCT07195565
Title: The Relationship Between Continuous Renal Replacement Therapy, Mortality, and Hospital Length of Stay in Critically Ill Burn Patients
Brief Title: Association of Continuous Renal Replacement Therapy With Mortality and Length of Stay in Critically Burned Patients
Acronym: CRRT-BURN
Status: Completed | Type: Observational
Sponsor: Pinar Timur Tasci (Other Government)
Responsible Party: Sponsor-Investigator, Pinar Timur Tasci, Resident Physician, Department of Anesthesiology and Reanimation, Dr. Lutfi Kirdar Kartal Training and Research Hospital
Organization: Dr. Lutfi Kirdar Kartal Training and Research Hospital (Other Government)
Other Study IDs: DrLutfiKirdarTRH-ANES-PTT-01
Record Dates: First submitted 2025-09-14; First posted 2025-09-26 (Actual); Last update posted 2025-09-26 (Actual); Status verified 2025-09

CONDITIONS: Severe Burns; Acute Kidney Injury; Critical Illness
Keywords: Continuous Renal Replacement Therapy; RIFLE Criteria; Mortality; Hospital Length of Stay; Mechanical Ventilation; İnotropic Support
MeSH Terms: conditions — Burns; Acute Kidney Injury; Critical Illness

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This retrospective observational study aims to investigate the clinical outcomes of critically ill burn patients who underwent continuous renal replacement therapy (CRRT). Primary endpoints include the evaluation of RIFLE criteria, timing of CRRT initiation, and overall survival. Secondary endpoints consist of comorbidity status, requirement for mechanical ventilation, inotropic support, and hospital length of stay among non-survivors.

DETAILED DESCRIPTION:
Severe burn injury is frequently complicated by acute kidney injury (AKI), which is associated with high morbidity and mortality in intensive care settings. Continuous renal replacement therapy (CRRT) is often required in this patient population; however, the prognostic factors influencing survival remain incompletely defined.

In this retrospective study, we analyzed critically ill burn patients who required CRRT. The primary outcomes were the RIFLE classification at the time of CRRT initiation, the timing of therapy initiation, and patient survival. The secondary outcomes included the presence of comorbidities, the need for mechanical ventilation, inotropic support, and length of hospital stay in non-survivors.

By systematically evaluating these clinical parameters, the study aims to clarify the prognostic impact of CRRT in burn patients and to contribute evidence for optimizing the management of acute kidney injury in this critically ill population.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged 18 years and older
* Admitted to and treated in the Burn Intensive Care Unit

Exclusion Criteria:

* Patients with an ICU stay of less than 24 hours
* Patients younger than 18 years
* Patients with known chronic kidney disease or history of kidney transplantation
* Patients admitted with toxic epidermal necrolysis (TEN)
* Patients with estimated glomerular filtration rate (eGFR) ≤ 15 mL/min/1.73m² at admission

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients (≥18 years) admitted to and treated in the Burn Intensive Care Unit.
Sampling Method: Non-Probability Sample
Enrollment: 238 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2024-01-01 (Actual); Study Completion 2024-01-01 (Actual)

PRIMARY OUTCOMES:
RIFLE criteria classification at CRRT initiation | Baseline( Day0, at CRRT initiation)
  Patients receiving CRRT will be classified according to the RIFLE criteria (Risk, Injury, Failure, Loss, End-stage kidney disease) at the time of CRRT initiation. The distribution across categories will be analyzed.
Timing of CRRT initiation | Baseline( Day0, at CRRT initiation, recorded from patient medical records)
  Date and time of initiation of continuous renal replacement therapy (CRRT), obtained from patient medical records.
Survival status of patients | At hospital discharge ( end of hospitalization)
  Survival versus non-survival status at the end of hospitalization.

SECONDARY OUTCOMES:
Presence of comorbidities in non-survivors | Baseline( Day0, at hospital admission)
  Documentation of chronic comorbidities (e.g., diabetes, hypertension, cardiovascular disease) in patients who died after CRRT.
Requirement for mechanical ventilation in non-survivors | Through ICU stay, up to hospital discharge (or death)
  Need for invasive mechanical ventilation among non-survivors receiving CRRT.
Requirement for inotropic support in non-survivors | Through ICU stay, up to hospital discharge or death
  Requirement for vasopressor or inotropic agents among non-survivors receiving CRRT.
Hospital length of stay in non-survivors | From hospital admission through study completion( up to discharge or death)
  Total length of hospitalization measured in days for patients who did not survive after CRRT.

CONTACTS AND LOCATIONS:
Overall Officials: Elif Bombaci, MD, Principal Investigator — Dr.Lutfi Kirdar City Hospital, Department of Anesthesiology and Reanimation, İstanbul, Turkey
Locations (1):
- Dr. Lutfi Kirdar City Hospital, Department of Anesthesiology and Reanimation, Istanbul, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
Individual participant data (IPD) will not be shared due to patient confidentiality and ethical considerations.